CLINICAL TRIAL: NCT03419975
Title: A Multi-center, Randomized,Blinded Evaluator, Active Control, Parallel, Phase III Study to Evaluate the Efficacy and Safety of TJO-002 in Primary Open Angle Glaucoma or Ocular Hypertension Patients
Brief Title: A Multi-center, Randomized, Blinded Evaluator, Active Control, Parallel, Phase III Study to Evaluate the Efficacy and Safety of TJO-002 in POAG or Ocular Hypertension Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Taejoon Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TJO-002-301
Record Dates: First submitted 2018-01-24; First posted 2018-02-05 (Actual); Last update posted 2019-09-04 (Actual); Status verified 2018-01

CONDITIONS: Primary Open-angle Glaucoma; Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — Latanoprost

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TJO-002 (Experimental)
  Interventions: Drug: TJO-002
- latanoprost (Active Comparator)
  Interventions: Drug: Latanoprost

INTERVENTIONS:
Drug: TJO-002 — Administrate the drugs for clinical trial one drop once daily at the same time (9 p.m. ± 1 hour) for a study eye
  Arms: TJO-002
Drug: Latanoprost — Administrate the drugs for clinical trial one drop once daily at the same time (9 p.m. ± 1 hour) for a study eye
  Arms: latanoprost

SUMMARY:
TJO-002 or Acitve Control was administered on primary open-angle glaucoma or ocular hypertension patients for 12 weeks. This clinical trial study has hypothesize TJO-002 administration groups are not inferior to Active control administration groups.

ELIGIBILITY:
* Inclusion Criteria:

  * Male or female, age 19 or over
  * Written informed consent to participate in the trial
* Exclusion Criteria:

  * Any other Galucoma except POAG(ex, Closed anterior chamber angle, angle-closure glaucoma)
  * Any laser or ocular surgery within 3months prior screening
  * Use of contact lenses
  * Known reactive airways disease
  * Any condition limiting patient's ability to participate in the trial

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Estimated)
Dates: Start 2016-04-26 (Actual); Primary Completion 2017-12-28 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
Change From Baseline in diurnal IOP at Week 12 | Baseline and Week 12
  After 12 weeks of administration of the drugs compare the therapeutic effectiveness between control drug and trial drug evaluated as the effect on reducing diurnal IOP.

SECONDARY OUTCOMES:
Change From Baseline in diurnal IOP at Week 8 | Baseline and Week 8
  After 8 weeks of administration of the drugs compare the therapeutic effectiveness between control drug and trial drug evaluated as the effect on reducing diurnal IOP.

CONTACTS AND LOCATIONS:
Locations (1):
- Chan Yun, Kim, Seoul, South Korea